CLINICAL TRIAL: NCT00245245
Title: An Open-Label Study of the Hemostatic Activity, Pharmacokinetics and Safety of OBI-1 (B-Domain Deleted Recombinant Porcine FVIII), When Administered by Intravenous Injection, to Control Non-Life and Non-Limb Threatening Bleeding Episodes in Congenital Hemophilia A Patients With an Inhibitor to Human FVIII
Brief Title: Study of Recombinant Porcine Factor VIII (FVIII) in Hemophilia and Inhibitors to FVIII
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Octagen Corporation (Industry)
Collaborators: Biomeasure Inc, Ipsen Group (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OBI-1 - 201; NIH Grant 2R44 HL064497-02
Record Dates: First submitted 2005-10-25; First posted 2005-10-27 (Estimated); Last update posted 2007-10-04 (Estimated); Status verified 2007-10

CONDITIONS: Hemophilia A
Keywords: hemophilia A; inhibitor; treatment
MeSH Terms: conditions — Hemophilia A | interventions — ZNF717 protein, human

INTERVENTIONS:
Drug: recombinant porcine coagulation factor VIII (OBI-1)

SUMMARY:
The ability of a new recombinant porcine coagulation factor VIII, B-domain deleted (called "OBI-1"), to control the non-life- or limb-threatening bleeding episodes patients with hemophilia A commonly develop is being evaluated. Patients with congenital hemophilia A and a low-titer (<20 Bethesda units [Bu]) inhibitory antibody to OBI-1, who meet the inclusion/exclusion criteria, will receive OBI-1 to treat their soft tissue or joint bleeding episode. At least the first two treatment episodes will be performed in the controlled setting of the hemophilia center/clinic/office, where any side effects can be observed. If the patient continues to meet the inclusion/exclusion criteria, has had no serious or severe adverse reactions to OBI-1, and has been in a home care program, the investigator may permit the patient to self-administer OBI-1 at home to treat subsequent bleeding episodes. The study will continue at least until 12 or more patients have received at least 24 treatment episodes in the aggregate.

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate the hemostatic activity of OBI-1 to control a bleeding episode in hemophilia A patients with inhibitors who are experiencing a non-life and/or non-limb threatening bleeding episode.

The secondary objectives of this study will be to assess the:

* safety of OBI-1,
* serial anti-OBI-1 and anti-human factor VIII (fVIII) inhibitor antibody responses following therapeutic administration of OBI-1, and
* pharmacokinetics of OBI-1 administered to control a bleeding episode.

After qualifying for the study at a Screening visit, patients will come to the investigator for treatment of a qualifying bleeding episode. After baseline blood samples are taken for inhibitor titer, a Loading Dose of OBI-1, calculated to inactivate the inhibitor, will be administered intravenously. After a blood sample is drawn to measure inhibitor titer and fVIII level, a Treatment Dose of 50 U/kg is administered. Serial blood samples will be drawn for fVIII levels for pharmacokinetics. At 6-hour intervals, additional Treatment doses, at increasing dose levels up to 150 U/kg, may be given if needed. Follow-up safety evaluations, beginning at Day 14, are scheduled; inhibitor titers against human fVIII and OBI-1 will be measured to assess continuing eligibility.

A second qualifying bleeding episode will be treated as the first, but without pharmacokinetic samples. If the patient's inhibitor titer against OBI-1 rises to > 20 Bu, further treatments with OBI-1 will be suspended until the titer decreases to 20 Bu or lower. Third and subsequent treatment episodes may be self-administered by the patient, under strict supervision of the investigator, in home care.

The study will continue until at least 12 patients have received at least 24 treatments, unless the Data Safety Monitoring Committee (DSMC) recommends a change in dosing calculations sooner.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet at least the following criteria to participate in the trial:

* Age at least 12 years.
* Clinical diagnosis of congenital hemophilia A with current inhibitor to human fVIII OR the patient is known to have developed an anti-human fVIII inhibitor antibody anamnestic response to human fVIII in the past.
* OBI-1 inhibitor antibody titer < 20 Bethesda Units at screening.
* Uncomplicated joint or soft tissue bleed, or other non-life threatening or non-limb threatening bleeding episode.

Exclusion Criteria:

Patients will be ineligible to participate if any of the following are present:

* Current treatment plan for any acute bleeding episode incorporates the use of human fVIII (recombinant or plasma-derived).
* Presence of any life- or limb-threatening bleeding episode (defined)
* Patient has received any human fVIII or prothrombin complex concentrate (PCC), within 7 days prior to Screening, OR received any PCC within 7 days prior to treatment with OBI-1.
* Patient has received recombinant human fVIIa (rVIIa) within 3 days prior to Screening OR within 3 days prior to treatment with OBI-1.
* Significant liver disease or renal disease

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2005-05; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
The percentage of successful treatment episodes, defined as having achieved control of the bleeding episode within One Loading Dose and 8 or fewer Treatment Doses, with a dose limit of 1000 U/kg in 24 hours

SECONDARY OUTCOMES:
Adverse events and serious adverse events observed throughout course of study
Pattern of inhibitory antibody response to OBI-1 following treatments
The percentage of patients who continue to qualify because their anti-OBI-1 titer remains at 20 Bu or less
Pharmacokinetics of OBI-1 when it is administered for treatment of a qualifying bleeding episode, in the absence of an inhibitory antibody to OBI-1

CONTACTS AND LOCATIONS:
Overall Officials: Josef N Mueksch, MD, MBA, Principal Investigator — Octagen Corporation
Locations (1):
- Octagen Corporation, Blue Bell, Pennsylvania, United States